CLINICAL TRIAL: NCT01566630
Title: An Adaptive Multicentre, Randomized, Partially Double-blind, Placebo-controlled Study to Assess the Safety, PK and PD/Efficacy of RLX030 in Women With Pre-eclampsia
Brief Title: Safety and Efficacy of RLX030 in Pregnant Women With Pre- Eclampsia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis terminated this study due to internal, strategic decisions.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRLX030A2205; 2011-001617-14 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Pre-eclampsia
Keywords: human recombinant RLX030; Pre-eclampsia; hemodynamics; Pharmacokinetics
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- RLX030 (Experimental): In part 1, within each cohort, two (2) patients per cohort will be treated open label with RLX030 and two (2) patients will be treated double blind with RLX030 as intravenous infusion for 72 hours. There will be 3 cohorts in part 1 with different doses of RLX030.
  In part 2, there is no open label treatment on RLX030. In part 2, patients will be randomized in a double-blind fashion to this arm with the optimal dose of RLX030 as intravenous infusion for 72 hours as determined from part 1.
  Interventions: Drug: RLX030
- Placebo (Placebo Comparator): In part 1, equal number of subjects will be treated with matching placebo of RLX030 as intravenous infusion for 72 hours in 3 cohorts.
  In part 2, patients will be treated with matching placebo of RLX030 as intravenous infusion for 72 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo to RLX030 as intravenous infusion for 72 hours
  Arms: Placebo
Drug: RLX030 — RLX030 1 mg/mL vials
  Arms: RLX030

SUMMARY:
This study is designed in two parts. Part 1 will assess the safety and tolerability of different doses of RLX030 when given to pregnant women with pre- eclampsia (elevated blood pressure with protein in urine). Part 2 will assess whether an optimal dose of RLX030 can prolong pregnancy in women with pre-eclampsia.

ELIGIBILITY:
Key Inclusion criteria:

* Written informed consent was obtained before any assessment was performed.
* Women at 18 to 40 years of age with a pregnancy 28 weeks (0 days) and 33 weeks (+4 days) gestational age. Gestational age was based on mother's last menstruation; if last menstruation was unknown, an alternative method was used as applicable and was documented in the (electronic) Case Report/Record Form [(e)CRF].
* Women with a diagnosis of pre-eclampsia or superimposed pre-eclampsia requiring hospitalization. Pre-eclampsia was defined as new onset of hypertension (SBP ≥ 140 or DBP ≥ 90 mmHg) or gestational hypertension accompanied by proteinuria (>= 0.3 g/24h) after 20 weeks of gestation. Superimposed pre-eclampsia was defined as chronic hypertension with new onset of proteinuria after 20 weeks of gestation.
* Reassuring fetal testing (cardiotocography and biophysical profile)

Key Exclusion criteria:

* Severe hypertension (SBP ≥ 160 mmHg or DBP ≥ 110 mmHg) and /or those receiving anti-hypertensive treatment at time of randomization.
* Clinically relevant electrocardiogram (ECG) abnormalities at screening excluding those abnormalities commonly seen in pregnancy according to the Investigator.
* Symptoms indicative of severe pre-eclampsia or HELLP syndrome (Hemolysis, Elevated Liver enzymes, and Low Platelet count) for which immediate delivery of the baby may be indicated. Symptoms include persistent CNS symptoms (severe headaches, visual changes, altered mentation), persistent right upper quadrant or epigastric pain, nausea or vomiting, severe thrombocytopenia (<100,000/mm3) and abnormal (> 2X upper limit of normal) liver enzymes (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]).
* Eclampsia during current pregnancy, vaginal bleeding present at screening, abruptio placentae, oligohydramnios
* Current diagnosis of a seizure disorder that requires chronic medication.
* Pre-gestational diabetes (Type 1 or Type 2) with or without diabetic retinopathy. Diagnosis (previous or current) of gestational diabetes, regardless of treatment, was allowed
* Known allergy to magnesium sulfate or steroids.
* Multifetal gestation, known major fetal anomaly, intrauterine growth restriction (<5th percentile).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (4):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Galveston, Texas
- Novartis Investigative Site, Modena, MO, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- RLX030: Because premature termination of the study, only Cohort 1 part 1 had patients with early onset pre-eclampsia. As per planned treatment assigned, patients in this arm received open label serelaxin (RLX030) 15 μg/kg/day i.v. for 72 hours.
- Placebo: Because premature termination of the study, only Cohort 1 part 1 had patients with early onset pre-eclampsia. The randomized patient received matching placebo of serelaxin (RLX030) in a blinded manner.
Period: Overall Study
Arm/Group | RLX030 | Placebo
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RLX030 | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Customized [Number; unit: Participants] — Between age 18 to 40
  Participants
    Between age 18 to 40 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events, Serious Adverse and Death During Part 1 of the Study
Description: Safety and tolerability was assessed by adverse events/serious adverse event and death monitoring.
Time Frame: Prior to delivery until 4-6 weeks post partum (maximum of 8 weeks)
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed.
Measure: Number; unit: Participants
Groups:
- RLX030 - Maternal: Because premature termination of the study, only Cohort 1 part 1 had patients with early onset pre-eclampsia. Serelaxin (RLX030) 15 μg/kg/day i.v. for 72 hours received by pregnant patients with early onset pre-eclampsia
- Placebo - Maternal: Because premature termination of the study, only Cohort 1 part 1 had patients with early onset pre-eclampsia. Matching placebo to serelaxin (RLX030) received for 72 hours by pregnant patients with early onset pre-eclampsia
- RLX030- Neonates Born to Patients: Neonates born to patients who received Serelaxin (RLX030) 15 μg/kg/day i.v. for 72 hours received
- Placebo- Neonates Born to Patients: Neonates born to patients who received placebo for 72 hours received by pregnant patients with early onset pre-eclampsia
Arm/Group | RLX030 - Maternal | Placebo - Maternal | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 2 | 1 | 2 | 1
Participants
  Serious Adverse events | 2 | 1 | 2 | 1
  Death | 0 | 0 | 0 | 0
  Non-serious AEs | 2 | 1 | 2 | 0

2. Primary Outcome: Change From Baseline in Maternal Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in Part 1of the Study (Part 1)
Description: Maternal safety assessment to monitor pre-eclampsia by checking blood pressure during 72 hour treatment period as well as post-dose.
Time Frame: From baseline to during treatment period of a maximum 72 hours infusion prior to delivery until 4-6 weeks post partum in part 1 (maximum of 8 weeks)
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change From Baseline in Mean Maternal Arterial Pressure (Part 1)
Description: Maternal safety assessment to monitor pre-eclampsia by checking mean arterial pressure during 72 hour treatment period as well as post-dose.
Time Frame: as for outcome 2
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change From Baseline on Maternal Proteinuria (Part 1)
Description: Pre-eclampsia was monitored by checking levels of protein in urine and by urinary protein/creatinine ratio (UPCR)
Time Frame: as for outcome 2
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Decrease in Utero-placental Blood Flow (Part 1)
Description: Blood flow to the fetus was monitored using via a Doppler.
Time Frame: During treatment period of a maximum 72 hours infusion prior to delivery and up to delivery in part 1 (maximum of 3 weeks)
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change in Fetal Heart Rate (Part 1)
Description: Heart rate of fetus was monitored continuously throughout 72 hour treatment period using a cardiotocograph.
Time Frame: as for outcome 5
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Improvement in Renal Function Assessed by Increase in Creatinine Clearance
Time Frame: From randomization until 4-6 weeks post partum (maximum 8 weeks)
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Rate of Spontaneous Delivery and/or Mode of Delivery
Time Frame: From randomization to delivery (maximum of 3 weeks)
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Number of Patients With Absence of Anti-serelaxin Antibodies
Time Frame: From Randomization until 4-6 weeks post partum (maximum of 8 weeks)
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Patients With Abnormalities in Birth Weight, Gestational Age, Appearance, Pulse, Grimace, Activity, Respiration (APGAR) Score, Umbilical Cord Gases, and Days in Neonatal Intensive Care Unit (NICU)
Time Frame: up to 4 - 6 weeks post partum (maximum of 8 weeks )
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Number of Patients With Abnormalities in Fetal Cardiotocography and Biophysical Profile
Time Frame: Randomization to delivery (maximum of 3 weeks)
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Pharmacokinetics of RLX030: Area Under the Blood Concentration-time Curve From Time Zero to Infinity (AUCinf)-Part 1
Description: Blood concentrations of RLX-030 was assayed to determine this PK parameter.
Time Frame: Baseline, 2, 6, 24,48,72, 76, 80 and 90 hours after initiation of infusion during part 1
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Primary Outcome: Pharmacokinetics of RLX030: Area Under the Blood Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast)-Part 1
Description: Blood concentrations of RLX-030 was assayed to determine this PK parameter.
Time Frame: Baseline, 2, 6, 24,48,72, 76, 80 and 90 hours after initiation of infusion during part 1
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Primary Outcome: Pharmacokinetics of RLX030: Blood Concentration at 24 Hour (C 0-24h) After Administration- Part 1
Description: Blood concentrations of RLX-030 was assayed to determine this PK parameter.
Time Frame: Baseline, 2, 6, 24,48,72, 76, 80 and 90 hours after initiation of infusion during part 1
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Primary Outcome: Pharmacokinetics of RLX030: Terminal Elimination Half-life (T1/2)- Part 1
Description: Blood concentrations of RLX-030 was assayed to determine this PK parameter.
Time Frame: Baseline, 2, 6, 24,48,72, 76, 80 and 90 hours after initiation of infusion during part 1
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Primary Outcome: Pharmacokinetics of RLX030: Mean Residence Time (MRT)
Description: Blood concentrations of RLX-030 was assayed to determine this PK parameter.
Time Frame: Baseline, 2, 6, 24,48,72, 76, 80 and 90 hours after initiation of infusion during part 1
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal | RLX030- Neonates Born to Patients | Placebo- Neonates Born to Patients
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Mean Number of Days Before Delivery
Time Frame: From randomization until delivery (maximum of 3 weeks)
Population: No formal analysis was performed as the study was terminated after three patients were enrolled and dosed
Arm/Group | RLX030 - Maternal | Placebo - Maternal
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The safety evaluation population included all patients who commenced study drug infusion. Safety reportied on all patients and their neonates.
Groups:
- RLX030- Maternal: Serelaxin (RLX030) 15 μg/kg/day i.v. for 72 hours received by pregnant patients with early onset pre-eclampsia
- Placebo- Maternal: Matching placebo to serelaxin (RLX030) received for 72 hours by pregnant patients with early onset pre-eclampsia
Arm/Group | RLX030- Maternal | RLX030- Neonates Born to Patients | Placebo- Maternal | Placebo- Neonates Born to Patients
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 1/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RLX030- Maternal (N=2) | RLX030- Neonates Born to Patients (N=2) | Placebo- Maternal (N=1) | Placebo- Neonates Born to Patients (N=1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 1
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 1 | 0
Caesarean section (Surgical and medical procedures) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RLX030- Maternal (N=2) | RLX030- Neonates Born to Patients (N=2) | Placebo- Maternal (N=1) | Placebo- Neonates Born to Patients (N=1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Mechanical ventilation (Surgical and medical procedures) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.